CLINICAL TRIAL: NCT07390539
Title: A Phase 1/1b Study of Autologous b7-h3 Chimeric Antigen Receptor t Cells (b7-h3.cd28z.Cart) in Children and Young Adults With Recurrent or Progressive Cns Neoplasms Expressing b7-h3 Target
Brief Title: B7-H3.CD28Z.CART in CNS Neoplasms
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Robbie Majzner (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Robbie Majzner, Sponsor-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25-642
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Central Nervous System Neoplasms; Brain Tumor; Brain Tumor, Recurrent; Brain Tumor, Pediatric; Brain Tumor Adult; Medulloblastoma; Medulloblastoma, Childhood; Medulloblastoma, Adult; Medulloblastoma Recurrent; Ependymoma; Atypical Teratoid/Rhabdoid Tumor; Embryonal Tumor With Multilayered Rosettes; Pineoblastoma; Leptomeningeal Disease
Keywords: Central Nervous System Neoplasms; Brain Tumor; Brain Tumor, Pediatric; Brain Tumor, Adult; Brain Tumor Recurrent; Medulloblastoma; Medulloblastoma, Childhood; Medulloblastoma, Adult; Medulloblastoma Recurrent; Ependymoma; Atypical Teratoid/Rhabdoid Tumor; Embryonal Tumor with Multilayered Rosettes; Pineoblastoma; Leptomeningeal Disease
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Medulloblastoma; Ependymoma; Rhabdoid Tumor; Neuroectodermal Tumors, Primitive; Pinealoma; Meningeal Neoplasms | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: dose-escalation by modified 3+3 in two risk strata, followed by dose expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation for B7-H3.CD28Z.CART in Standard Risk Stratum (Experimental): Participants will be enrolled in a staggered, sequential fashion using a modified 3 + 3 dose escalation design, assigning participants to one of three intravenous dose levels to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of IV B7-H3.CD28Z.CART. Dose escalation will occur per dose-limiting toxicity rules.
  * Baseline visit
  * Apheresis to obtain T cells
  * Days -4, -3, -2: predetermined doses of Fludarabine and Cyclophosphamide 1x daily
  * Day 0: B7-H3 CAR T cell infusion 1x daily
  * 2 doses of B7-H3 CAR T cell infusion Intracerebroventricular (ICV) Infusion every 28 days until 8 doses total according to clinical response
  * Follow up every 3 months after last infusion up until 2 years
  * Long term follow annually for an additional 13 years
  Interventions: Biological: B7-H3.CD28Z.CART; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Escalation for B7-H3.CD28Z.CART in High Risk Stratum (Experimental): Participants will be enrolled in a staggered, sequential fashion using a modified 3 + 3 dose escalation design, assigning participants to one of three intravenous dose levels to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of IV B7-H3.CD28Z.CART. Dose escalation will occur per dose-limiting toxicity rules.
  * Baseline visit
  * Apheresis to obtain T cells
  * Days -4, -3, -2: predetermined doses of Fludarabine and Cyclophosphamide 1x daily
  * Day 0: B7-H3 CAR T cell infusion 1x daily
  * 2 doses of B7-H3 CAR T cell infusion Intracerebroventricular (ICV) Infusion every 28 days until 8 doses total according to clinical response
  * Follow up every 3 months after last infusion up until 2 years
  * Long term follow annually for an additional 13 years
  Interventions: Biological: B7-H3.CD28Z.CART; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Expansion for B7-H3.CD28Z.CART in Standard Risk Stratum (Experimental): Dose expansion will occur per dose-limiting toxicity rules.
  * Baseline visit
  * Apheresis to obtain T cells
  * Days -4, -3, -2: predetermined doses of Fludarabine and Cyclophosphamide 1x daily
  * Day 0: B7-H3 CAR T cell infusion 1x daily
  * 2 doses of B7-H3 CAR T cell infusion Intracerebroventricular (ICV) Infusion every 28 days until 8 doses total according to clinical response
  * Follow up every 3 months after last infusion up until 2 years
  * Long term follow annually for an additional 13 years
  Interventions: Biological: B7-H3.CD28Z.CART; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Expansion for B7-H3.CD28Z.CART in High Risk Stratum (Experimental): Dose expansion will occur per dose-limiting toxicity rules.
  * Baseline visit
  * Apheresis to obtain T cells
  * Days -4, -3, -2: predetermined doses of Fludarabine and Cyclophosphamide 1x daily
  * Day 0: B7-H3 CAR T cell infusion 1x daily
  * 2 doses of B7-H3 CAR T cell infusion Intracerebroventricular (ICV) Infusion every 28 days until 8 doses total according to clinical response
  * Follow up every 3 months after last infusion up until 2 years
  * Long term follow annually for an additional 13 years
  Interventions: Biological: B7-H3.CD28Z.CART; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: B7-H3.CD28Z.CART — Autologous CAR T cells targeting B7-H3 (CD276), administered intravenously (into the vein) per protocol.
Drug: Fludarabine — Lymphodepleting chemotherapy administered intravenously per institutional standards.
Drug: Cyclophosphamide — Lymphodepleting chemotherapy administered intravenously per institutional standards.

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of a cell therapy at different doses for children and young adults with recurrent or progressive brain tumors. Recurrent/recurred means a tumor that has gone away and then came back. This cell therapy is called B7- H3.CD28Z.CART, referred to as B7-H3 CAR T cells. B7-H3 is a protein that is over-expressed on many tumor cells, making it a good target for cancer cell therapy.

The names of the study investigational therapies involved in this study are:

* Fludarabine (a type of chemotherapy)
* Cyclophosphamide (a type of chemotherapy)
* B7-H3 CAR T cells (a type of cellular therapy)

DETAILED DESCRIPTION:
This is a single-institution, Phase 1/1b, open-label study to test the safety and effectiveness of a cell therapy at different doses for children and young adults with recurrent or progressive brain tumors. Recurrent/recurred means a tumor that has gone away and then came back. This cell therapy is called B7- H3.CD28Z.CART, referred to as B7-H3 CAR T cells. B7-H3 is a protein that is over-expressed on many tumor cells, making it a good target for cancer cell therapy.

The U.S. Food and Drug Administration (FDA) has not approved B7-H3 CAR T cells as a treatment for any disease.

Fludarabine and cyclophosphamide are standard lymphodepleting chemotherapy medications that are being used in this study to prepare the body for cell therapy. They are approved by the U.S. Food & Drug Administration (FDA) for this purpose and are not intended to be treatment for recurrent or progressive brain tumors.

The structure of the study will be by dose-escalation using a modified 3+3 design in two risk strata (standard risk, high risk), followed by a two-stage Phase 1b expansion at the recommended Phase 2 dose.

Participation in this study is expected to last up to 15 years.

It is expected that about 70 people will participate in this study.

ELIGIBILITY:
Pre-screening Inclusion Criteria:

* Participants must have histologically and/or molecularly confirmed CNS embryonal tumor (see eligible tumor types below), OR ependymoma that is recurrent/progressive following standard of care treatment.

  --Eligible CNS embryonal tumor types include:
  * Medulloblastoma
  * Atypical Teratoid Rhabdoid Tumor (ATRT)
  * Embryonal Tumor with Multilayered Rosettes (ETMR) Pineoblastoma
  * Other CNS embryonal tumor types, at the discretion of the study chair (or designee)
* Participants must have adequate pre-trial tumor material available to determine B7- H3 expression status. Tumor tissue from the most recent resection or biopsy of recurrent disease is preferred. If unavailable, tumor tissue from prior recurrences or from time of initial diagnosis is acceptable. Biopsies will not be performed for participation in this research trial or for research purposes.
* Pre-screening IHC Consent: All participants ≥ 18 years of age must be able to give informed consent. For participants <18 years of age, their legal authorized representative (LAR) (i.e. parent or guardian) must give informed consent. Pediatric participants will be included in age-appropriate discussion and written assent will be obtained for those ≥10 years of age, where appropriate. If a minor becomes of age during participation of this study, they will be asked to reconsent as an adult.

Inclusion Criteria:

* Participants must have histologically and/or molecularly confirmed CNS embryonal tumor (see eligible tumor types below), OR ependymoma that is recurrent/progressive following standard of care treatment.

  --Eligible CNS embryonal tumor types include:
  * Medulloblastoma
  * Atypical Teratoid Rhabdoid Tumor (ATRT)
  * Embryonal Tumor with Multilayered Rosettes (ETMR)
  * Pineoblastoma
  * Other CNS embryonal tumor types, at the discretion of the study chair (or designee)
* B7-H3 expression: Demonstration of B7-H3 expression with H score greater than 100 by immunohistochemistry (IHC) is required.
* Age: greater than or equal to two (2) years of age and less than or equal to 21 years of age. The first participant treated at each dose level within each stratum (Standard Risk and High Risk) will be ≥ 6 years of age when feasible.
* Disease status: Participants must have evaluable disease in the central nervous system to be eligible. Evaluable disease includes either measurable OR non-measurable disease, defined as follows:

  --Measurable disease (contrast-enhancing or non-enhancing tumor)
  * Clearly defined lesional margins with two perpendicular diameters of at least 10mm, OR
  * At least two times (in both perpendicular diameters) the MRI slice thickness, plus the interslice gap

    --Non-measurable disease (tumor that is too small to be accurately measured)
  * Lesion that is measurable in only one perpendicular dimension, OR
  * Lesion that is less than 10mm in at least one perpendicular dimension, OR
  * Lesion that is less than two times the MRI slice thickness, plus the interslice gap
  * Note: Leptomeningeal (LM) disease is considered non-measurable but evaluable.
* Performance status: Karnofsky performance status ≥60% for participants ≥16 years of age and Lansky performance status ≥60% for participants <16 years of age (see APPENDIX A PERFORMANCE STATUS CRITERIA). NOTE: Participants with neurologic deficits must have a stable neurologic exam for seven (7) days prior to enrollment. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Life expectancy of greater than 12 weeks
* Prior therapy: Participants must have received prior standard of care therapy, including maximal safe surgical resection, radiation therapy and/or standard chemotherapy, and is recovered from all acute treatment-related toxicities (defined as ≤ Grade 1 or stable) from all prior therapy before entering this study There is no upper limit to the number of prior therapies allowed, but must have received all standard curative options for their tumor type.
* Participants must meet the following washouts prior to enrollment:

  * Radiation therapy - Participants must have had their last fraction of:

    ---Craniospinal irradiation, whole brain radiation therapy, or radiation therapy to >50% of the pelvis or spine >28 days prior to enrollment

    ---Focal irradiation (small port) >14 days prior to enrollment
  * At least 14 days since any prior cytotoxic chemotherapy
  * At least 7 days since any biologic antineoplastics, tyrosine kinase inhibitor, targeted agent
  * At least 21 days or 5 half-lives (whichever is shorter) since any investigational antineoplastic or disease-directed agent (but at least 28 days from prior investigational antineoplastic vaccine therapy)
  * At least 21 days since any monoclonal antibody therapy
  * At least 90 days since any systemic inhibitor/stimulatory immune checkpoint therapy
  * At least 28 days from prior autologous stem cell transplantation, with no ongoing toxicities
  * At least 14 days after peg-filgrastim and 7 days for hematopoietic growth factor support
* Steroid use: Must not require concurrent systemic steroid therapy, although physiologic corticosteroid replacement therapy for management of pituitary/adrenal insufficiency and/or topical administration (e.g. inhaled or dermatologic) is allowed. Use of topical, ocular, intranasal, or inhaled corticosteroids are permitted per PI

discretion.

* Participants must have adequate organ function, as defined below

  --Adequate bone marrow function
  * Hemoglobin ≥ 8 g/dL
  * Absolute neutrophil count (ANC) ≥ 1000 cells/uL
  * Absolute lymphocyte count (ALC) ≥ 150 cells/uL
  * Platelets ≥100,000/uL (unsupported, defined as no platelet transfusion within 4 days)
* Adequate renal function defined as creatinine within normal limits for age OR creatinine clearance (as estimated by Cockcroft Gault Equation for participants ≥ 18yo and Bedside Schwartz for participants <18yo) ≥70mL/min

  * Maximum Serum Creatinine mg/DL ---6 months to 1 year Male 0.5 Female 0.5 ---1 to < 2 years Male 0.6 Female 0.6 ---2 to < 6 years Male 0.8 Female 0.8

    * 6 to < 10 years Male 1 Female 1
    * 10 to < 13 years Male 1.2 Female 1.2
    * 13 years to < 16 years Male 1.5 Female 1.4

      * 16 years Male 1.7 Female 1.4
* Adequate hepatic function

  * Serum ALT/AST ≤3.0 upper limit of normal (ULN)
  * Total bilirubin ≤1.5mg/dL, except in subjects with confirmed Gilbert's syndrome
* Adequate cardiac function

  --Ejection fraction ≥50% or fractional shortening ≥28%, measured by echocardiography
* Adequate pulmonary function

  * No evidence of dyspnea at rest
  * Pulse oximetry >92% whilst breathing room air
* Adequate neurologic function

  * Participants with seizure disorders on anticonvulsants may be enrolled if seizures are well controlled (no seizure activity within 7 days prior to enrollment)
  * Nervous system disorders (CTCAE v6.0) resulting from prior therapy must be ≤ Grade 2, with the exception of decreased tendon reflex (DTR; any Grade eligible). Participants with neurological deficits should be stable for a minimum of 7 days prior to enrollment. (A baseline detailed neurological exam should clearly document the neurological status of the participant prior at enrollment).
* Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization are not considered to be of childbearing potential)
* Participants of childbearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for one year after receiving the preparative lymphodepletion regimen, or for as long as B7- H3.CD28Z.CART cells are detectable in peripheral blood or CSF, whichever is later.
* Participant or parent of participant or legally recognized representative must be able to sign a written informed consent document. Pediatric participants will be included in age-appropriate discussion and written assent will be obtained for those ≥10 years of age, where appropriate.

Exclusion Criteria:

* Participants with bulky tumor are ineligible. Bulky tumor is defined as:

  * Tumor with diameter of >5cm in one dimension on T2/FLAIR sequence
  * Tumor with evidence of clinically significant midline shift or uncal herniation
  * Tumor that, in opinion of the site investigator, shows significant mass effect in either the brain or spine
* Participants with clinical or radiological evidence of brain herniation.
* Participants who have received other B7-H3 targeted cellular therapies. Other prior cellular therapies are eligible, including immune checkpoint inhibition and vaccine therapy. These prior therapies should be discussed with the study chair (or designee) prior to participant enrollment.
* Concurrent illness

  * Participants with any prior immunodeficiency or history of autoimmune disease requiring systemic steroids/ immunosuppressive medication/ disease-modifying agents within the last two (2) years.
  * Uncontrolled (Grade 3) bacterial, viral, fungal, or other infection.
  * Ongoing infection with HIV or hepatitis B (HBsAg positive) or hepatitis C virus (anti-HCV positive). A history of hepatitis B or hepatitis C is permitted if the viral load is undetectable per quantitative PCR and/or nucleic acid testing.
  * Evidence of severe or uncontrolled systemic disease (e.g. Grade 3 significant cardiac, pulmonary, hepatic, renal or other organ dysfunction) that in the judgement of the principal investigator is likely to interfere with assessment of safety or efficacy of the investigational regimen and its requirements.
  * Known sensitivity or allergy to any of the agents/reagents used in this study (i.e. DSMO, cyclophosphamide, fludarabine)
  * History of severe hypersensitivity reaction to compounds of similar chemical or biologic compositions to any agent used in the study or in the manufacturing of cells.
* Concomitant medications

  * Current systemic corticosteroid therapy
  * Note, physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency will be allowed.
  * Participants who are receiving any other anti-cancer or investigational drug therapy are ineligible.
  * Participants who have received the last vaccination of a live vaccine ≤ 30 days prior to the start of treatment are ineligible.
  * Ongoing use of dietary supplements, alternative therapies or extreme diets, or any medication not approved by the study chair (or designee).
* Any other condition which in the principal investigator's opinion makes the individual clinically unsuitable to participate in this trial, or which would jeopardize compliance with the protocol, or would make it difficult to interpret adverse events or study data.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2030-08-31 (Estimated); Study Completion 2032-08-31 (Estimated)

PRIMARY OUTCOMES:
Manufacturing Success Rate of Autologous B7-H3.CD28Z CAR T Cells | Participants will receive the CART cell infusion on Day 0.
  Each participant's product will be tested for the following criteria: cell viability ≥ 70%; cell number within ± 20% of the planned dose; CD3+ T cells ≥ 80% of leukocytes; CAR-positive cells ≥ 10% of CD3+ T cells; endotoxin ≤ 5 EU/kg; mycoplasma not detected; vector copy number (VCN) per transduced cell ≤ 10; replication-competent retrovirus (RCR) not detected; and sterility confirmed as "No Growth to Date" (NGTD) after a minimum of 5 days in culture. A participant will be classified as a manufacturing success if the final product satisfies all release criteria. If any criterion is not met, the participant will be classified as a manufacturing failure. The manufacturing success rate is defined as the proportion of participants classified as a success.
Maximum Tolerated Dose (MTD) of B7-H3.CD28Z.CART Cells | 28 days
  The MTD is defined as the highest dose level of B7-H3.CD28Z.CART cells at which the rate of dose-limiting toxicity (DLT) is considered acceptable according to the modified 3+3 rules. Additional details are provided in Protocol Section 13.1. Definition of DLT is outlined in protocol. The definition of DLT uses NCI's Common Terminology Criteria for Adverse Events (CTCAEv6.0).
Recommended Phase 2 Dose (RP2D) of B7-H3.CD28Z.CART Cells | 28 days
  The recommended phase 2 dose (RP2D) is the dose of B7-H3.CD28Z.CAR T cells selected for Phase 2 based on Phase 1 results, considering safety, tolerability, manufacturing feasibility, and observed clinical activity, and may be at or below the Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD).

SECONDARY OUTCOMES:
Number of Participants Experience Dose-Limiting Toxicity (DLT) during Dose Escalation | 28 years
  Definition of DLT is outlined in protocol. The definition of DLT uses NCI's Common Terminology Criteria for Adverse Events (CTCAEv6.0).
Number of Participants Experience Dose-Limiting Toxicity (DLT) at Maximum Tolerated Dose (MTD) / Recommend Phase 2 Dose (RP2D) | 28 days
  Definition of DLT is outlined in protocol. The definition of DLT uses NCI's Common Terminology Criteria for Adverse Events (CTCAEv6.0).
Number of Participants with Two Additional ICV B7-H3.CD28Z.CAR T Infusions | From Day 0 (initial IV infusion) through Day 56 (third ICV infusion)
  The number of participants in the High-Risk Stratum who receive two additional intracerebroventricular (ICV) infusions of B7-H3.CD28Z.CAR T cells following the initial intravenous(IV) infusion.
Adverse Events of Special Interest (AESIs) Rate | From Day 0 (initial IV infusion) through Day 56 (third ICV infusion) plus a 28-day follow-up period, for a total of 74 days.
  AESIs rate is defined as the proportion of participants who experience AESIs during treatment period. AESIs is defined in protocol section 7.3. Adverse events will be summarized and graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 6.0.
Complete Response Rate (CRR) at Day 28 | Day 28
  CRR is defined as the proportion of participants who achieve complete response (CR) assessed by Response Assessment in Pediatric Neuro-Oncology (RAPNO) response guidelines for medulloblastoma and ependymoma. Immune-related response criteria (irRC) as defined in RANO 2.0 may be used to interpret responses potentially influenced by immune effects.
Partial Response Rate (PRR) at Day 28 | Day 28
  PRR is defined as the proportion of participants who achieve partial response (PR) assessed by Response Assessment in Pediatric Neuro-Oncology (RAPNO) response guidelines for medulloblastoma and ependymoma. Immune-related response criteria (irRC) as defined in RANO 2.0 may be used to interpret responses potentially influenced by immune effects.
Stable Disease Rate (SDR) at Day 28 | Day 28
  SDR is defined as the proportion of participants who achieve stable disease (SD) assessed by Response Assessment in Pediatric Neuro-Oncology (RAPNO) response guidelines for medulloblastoma and ependymoma. Immune-related response criteria (irRC) as defined in RANO 2.0 may be used to interpret responses potentially influenced by immune effects.
3 Month Complete Response Rate (CRR3) | 3 months
  CRR3 is defined as the proportion of participants who achieve complete response (CR) at 3 months, which assessed by Response Assessment in Pediatric Neuro-Oncology (RAPNO) response guidelines for medulloblastoma and ependymoma. Immune-related response criteria (irRC) as defined in RANO 2.0 may be used to interpret responses potentially influenced by immune effects.
3 Month Partial Response Rate (PRR3) | 3 months
  PRR3 is defined as the proportion of participants who achieve partial response (PR) at 3 months, which assessed by Response Assessment in Pediatric Neuro-Oncology (RAPNO) response guidelines for medulloblastoma and ependymoma. Immune-related response criteria (irRC) as defined in RANO 2.0 may be used to interpret responses potentially influenced by immune effects.
3 Month Stable Disease Rate (SDR3) | 3 months
  SDR3 is defined as the proportion of participants who achieve stable disease (SD) at 3 months, which assessed by Response Assessment in Pediatric Neuro-Oncology (RAPNO) response guidelines for medulloblastoma and ependymoma. Immune-related response criteria (irRC) as defined in RANO 2.0 may be used to interpret responses potentially influenced by immune effects.
Best Overall Response Rate (BORR) | Treatment duration may be up to 224 days, and disease evaluations will be performed at Day 28 (±4 days), at Months 2 and 3 (±1 week), and every 3 months thereafter through Month 24 (±4 weeks) after the end of treatment.
  BORR is defined as the proportion of participants who achieve a best overall response of complete response (CR), partial response (PR), or stable disease (SD) from the start of treatment until progressive disease (PD) or recurrence, taking as reference for progression the smallest measurements recorded since treatment initiation. Per Pediatric Neuro-Oncology (RAPNO) response guidelines, PD is defined as meeting any of the following criteria: a ≥25% increase in the sum of perpendicular diameters of measurable lesions or clear progression of non-measurable disease on MRI (brain/spine), appearance of any new lesion (biopsy confirmation if feasible), conversion of CSF cytology from negative to positive, clinical deterioration not attributable to other causes, or new extra-CNS disease.
Median Duration of Response (DOR) | Treatment duration may be up to 224 days, and disease evaluations will be performed at Day 28 (±4 days), at Months 2 and 3 (±1 week), and every 3 months thereafter through Month 24 (±4 weeks) after the end of treatment.
  DOR, estimated using the Kaplan-Meier method, is measured from the time when the criteria for complete response (CR) or partial response (PR) are first met until the first documented date of recurrent or progressive disease (PD) or death from any cause, using as reference for progression the smallest measurements recorded since treatment initiation. Participants without events are censored at the date of their last disease evaluation. Per Pediatric Neuro-Oncology (RAPNO) response guidelines, PD is defined as meeting any of the following criteria: a ≥25% increase in the sum of perpendicular diameters of measurable lesions or clear progression of non-measurable disease on MRI (brain/spine), appearance of any new lesion (biopsy confirmation if feasible), conversion of CSF cytology from negative to positive, clinical deterioration not attributable to other causes, or new extra-CNS disease.
2 Year Progression-Free Survival (PFS2) | 2 years
  PFS2 is the percent probability estimate at 2 years based on the Kaplan-Meier method. PFS is defined as the time from infusion of B7-H3.CD28Z.CART to the first occurrence of an event (progression, relapse, or death due to any cause). Participants alive without an event are censored at date of last disease evaluation. Per Pediatric Neuro-Oncology (RAPNO) response guidelines, PD is defined as meeting any of the following criteria: a ≥25% increase in the sum of perpendicular diameters of measurable lesions or clear progression of non-measurable disease on MRI (brain/spine), appearance of any new lesion (biopsy confirmation if feasible), conversion of CSF cytology from negative to positive, clinical deterioration not attributable to other causes, or new extra-CNS disease.
Median Overall Survival (OS) | 15 years
  OS based on Kaplan-Meier method is defined as the time from infusion of B7-H3.CD28Z.CART to death due to any cause, or censored at date last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Chi, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu